CLINICAL TRIAL: NCT06381713
Title: Short and Long Term Effect and Cost-utility of High Intensity vs. Low Intensity Speech Intervention in Children With Cleft Palate
Brief Title: Effect and Cost-utility of of High Intensity vs. Low Intensity Speech Intervention in Children With Cleft Palate
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: Research Foundation Flanders (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ONZ-2024-0158
Record Dates: First submitted 2024-04-08; First posted 2024-04-24 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Cleft Palate Children; Speech Therapy; Speech Disorders in Children; Cleft Lip and Palate
Keywords: Randomized controlled trial; Speech therapy; Cleft lip and palate
MeSH Terms: conditions — Communication Disorders; Cleft Lip

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High intensive speech therapy (Experimental): To investigate the (cost-)effectiveness of speech therapy for children with a cleft palate (with of without a cleft lip), we will provide a high-intensive speech intervention.
  Interventions: Behavioral: High intensive combined phonetic-phonological intervention
- Low intensive speech therapy (Active Comparator): To investigate the (cost-)effectiveness of speech therapy for children with a cleft palate (with of without a cleft lip), we will provide a low-intensive speech intervention.
  Interventions: Behavioral: Low intensive combined phonetic-phonological intervention

INTERVENTIONS:
Behavioral: High intensive combined phonetic-phonological intervention — Children will receive phonetic articulation therapy supplemented by phonological principles. Consonants will be treated with emphasis on phonetic placement and shaping techniques. Phonetic articulation therapy includes five different steps:(1) identification of the target consonant using visual, tactile, and auditory feedback techniques,(2) discrimination between the used and targeted consonant, (3) variation and correction, (4) stabilize the target, and (5) maintenance of the target. A next level will be introduced when the child is able to correctly produce the sound in 80% of the time with minimal cues from the therapist. Multiple errors will be targeted simultaneously by focusing on a process. Child-friendly games will be played to illustrate the contrast between concepts, for example glottal 'throat' sounds and oral 'mouth' sounds. Exercises will be embedded in meaningful language contexts such as minimal pairs.
  Therapy will be provided 5 times 30' per week for 2 times 4 weeks.
  Arms: High intensive speech therapy
Behavioral: Low intensive combined phonetic-phonological intervention — Children will receive phonetic articulation therapy supplemented by phonological principles. Consonants will be treated with emphasis on phonetic placement and shaping techniques. Phonetic articulation therapy includes five different steps:(1) identification of the target consonant using visual, tactile, and auditory feedback techniques,(2) discrimination between the used and targeted consonant, (3) variation and correction, (4) stabilize the target, and (5) maintenance of the target. A next level will be introduced when the child is able to correctly produce the sound in 80% of the time with minimal cues from the therapist. Multiple errors will be targeted simultaneously by focusing on a process. Child-friendly games will be played to illustrate the contrast between concepts, for example glottal 'throat' sounds and oral 'mouth' sounds. Exercises will be embedded in meaningful language contexts such as minimal pairs.
  Therapy will be provided 2 times 30' per week for 20 weeks.
  Arms: Low intensive speech therapy

SUMMARY:
Achieving speech that is understandable and acceptable to others is the key outcome in cleft treatment. Therefore, speech therapy provided by a speech-language pathologist is necessary. This intervention is traditionally provided twice per week for 30 minutes for months or even years by first-line speech-language pathologists. Unfortunately, this low intensity intervention is based on a historical context rather than scientific evidence. This means that current speech therapy knows several shortcomings including poor outcomes, treatment fatigue and high costs related to year-long therapy. Because of these issues, the use of high intensity speech intervention is proposed. Even though solid proof-of-concepts exist for this model, it has not yet found its way into clinical practice.

Before this intensity can be implemented and utilized in clinical practice, the effect of this novel program on a larger societal scale must be determined. This project will compare the effect of high intensity and low intensity speech intervention in children with a cleft palate in terms of speech, quality of life, and cost-utility as provided by first-line speech-language pathologists by conducting a large-scale randomized controlled trial. The final goal is to utilize this program in clinical practice and to create awareness of the benefits for children with a cleft palate among stakeholders.

DETAILED DESCRIPTION:
Objective 1: Conduct a large-scale randomized controlled trial to compare the short- and long-term sustainable effects of two different speech intervention intensities (i.e. high intensity speech intervention: 5x30 min/week during 2x4 weeks (2x10 hours) and low intensity speech intervention: 2x30 min/week during 20 weeks (20 hours)) on the speech and quality of life in Belgian Dutch-speaking children with a cleft palate with or without a cleft lip. Speech intervention will be provided by first-line speech language pathologists in private practices who will receive thorough training before the onset of the trial.

Hypothesis 1: Based on the state-of-the-art and our proof-of-concept, it is assumed that 20 hours of high intensity speech intervention will lead to superior speech outcomes and health-related quality of life compared to 20 hours of low intensity speech intervention.

Objective 2: To compare the cost-utility in quality-adjusted life years of two different speech intervention intensities (i.e. high intensity speech intervention: 5x30 min/week during 2x4 weeks (2x10 hours) and low intensity speech intervention: 2x30 min/week during 20 weeks (20 hours)) in Belgian Dutch-speaking children with a cleft palate with or without a cleft lip. Demonstrating the cost-effectiveness of high intensity speech intervention will facilitate implementation and utilization of this protocol in clinical practice as less money has to be spent in order to gain one life year in full health (QALY) when providing high intensity speech intervention compared to low intensity speech intervention.

Hypothesis 2: Besides the superior speech outcomes and health related quality of life in a shorter intervention time (cfr. hypothesis 1), it is hypothesized that less money has to be spent in order to gain one life year in full health (QALY) in the high intensity intervention group. In other words, it is hypothesized that high intensity intervention will be more cost-effective compared to low intensity speech intervention.

ELIGIBILITY:
Inclusion Criteria:

* Belgian Dutch-speaking children with a cleft palate with or without a cleft lip
* Aged between 4 and 12 years,
* Presence of at least one compensatory speech error in their speech based on the perceptual assessment of one experienced speech-language pathologist

Exclusion Criteria:

* Children with syndromic clefts
* Oronasal fistula
* Velopharyngeal insufficiency
* Hearing disabilities based on pure tone audiometry (>25 dB HL)
* Cognitive and/or related learning disabilities or neuromuscular disorders

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2024-11-26 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Consonant proficiency | Assessment 2 weeks pre-intervention, immediately pre-intervention, after 10 hours of therapy, after a 12-week rest period, immediately post-intervention, at 1 week post-intervention, at 2 weeks post-intervention, at 3 months post-intervention
  Consonant proficiency will be measured in terms of percentage correctly produced consonants (%)
Incremental cost-utility ratio | After a 12-week rest period (high intensity arm), at 3 months post-intervention
  The cost-utility of the high intensity speech intervention compared to the low intensity speech intervention will be examined by calculating the ratio of the incremental costs to the incremental health effects (QALYs) called the incremental cost-utility ratio (ICUR), calculated as Cost intervention - Cost control / Effect intervention - Effect control.
  The EQ-5D-Youth version will be used for children aged 8-12 years and the EQ-5D proxy version for children aged 4-7 years to collect information on HRQoL ("utilities").
  Cost information will be obtained using a self-reported questionnaire on health care use.
Incremental cost-effectiveness ratio | After a 12-week rest period (high intensity arm), at 3 months post-intervention
  The cost-effectiveness of the high intensity speech intervention compared to the low intensity speech intervention will be examined by calculating the ratio of the incremental costs to the incremental health effects (percentage correctly produced consonants) called the incremental cost-effectiveness ratio (ICER), calculated as Cost intervention - Cost control / Effect intervention - Effect control.
  The effectiveness will be estimated using the primary outcome (percentage correctly produced consonants) obtained from the randomized controlled trial.
  Cost information will be obtained using a self-reported questionnaire on health care use.

SECONDARY OUTCOMES:
Intelligibility in Context | Assessment immediately pre-intervention, after 10 hours of therapy, after a 12-week rest period, immediately post-intervention, at 3 months post-intervention
  To assess possible transfer of learned speech skills to contexts outside the therapy setting, the Intelligibility in Context Scale (ICS) will be administered. The ICS rates the degree to which children's speech is understood by different partners (caregivers, immediate and extended family, friends, acquaintances, teachers, and strangers) on a 5-point scale (1 - never intelligible to 5 - always intelligible)
Health-related quality of life | Assessment immediately pre-intervention, after 10 hours of therapy, after a 12-week rest period, immediately post-intervention, at 3 months post-intervention
  To evaluate the psychosocial impact of the interventions, the Velopharyngeal insufficiency Effects on Life outcomes (VELO) questionnaire will be administered. This tool consists of a caregiver and child report (for children older than 8 years) addressing different domains: speech limitation, swallowing problems, situational difficulty, emotional impact, perception by others, and caregiver impact. The higher the score, the better the health related quality of life.
Speech Function | Assessment immediately pre-intervention, after 10 hours of therapy, after a 12-week rest period, immediately post-intervention, at 3 months post-intervention
  The subscale "Speech Function" from the Dutch CLEFT-Q will be administered to measure how often someone has trouble speaking. This scale consists of 10 questions. Scores range from 0 to 100. Higher scores indicate less trouble speaking. This scale was developed and validated for children with CP±L between 8 and 29 years of age. Consequently, this scale will only be administered to children aged 8 years and older.
Speech Distress | Assessment immediately pre-intervention, after 10 hours of therapy, after a 12-week rest period, immediately post-intervention, at 3 months post-intervention
  The subscale "Speech Distress" from the Dutch CLEFT-Q will be administered to assess in more detail the feelings someone has regarding speaking. This scale consists of 10 questions. Scores range from 0 to 100. Higher scores indicate less negative feelings. This scale was developed and validated for children with CP±L between 8 and 29 years of age. Consequently, this questionnaire will only be administered to children aged 8 years and older.
Communication attitudes of children aged 4 and 5 years | Assessment immediately pre-intervention, after 10 hours of therapy, after a 12-week rest period, immediately post-intervention, at 3 months post-intervention
  To evaluate the change in communication attitudes of children aged 4 and 5 years during the intervention, the KiddyCAT will be administered before, during and after the intervention. This questionnaire evaluates the extent to which the child has a negative attitude toward speaking.
  The higher the score, the more negative the attitude toward speaking. the scores range from 0 (no negative communication attitudes) to 14 (negative communication attitudes only).
Communication attitudes of children aged 6 years and older | Assessment immediately pre-intervention, after 10 hours of therapy, after a 12-week rest period, immediately post-intervention, at 3 months post-intervention
  To evaluate the change in communication attitudes of children aged 6 years and older during the intervention, the Communication Attitudes Test (CAT) will be administered before, during and after the intervention. This questionnaire evaluate the extent to which the child has a negative attitude toward speaking.
  The higher the score, the more negative the attitude toward speaking. the scores range from 0 (no negative communication attitudes) to 33 (negative communication attitudes only).

CONTACTS AND LOCATIONS:
Overall Officials: Kristiane Van Lierde, PhD, Principal Investigator — University Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No